CLINICAL TRIAL: NCT07292961
Title: Investigating the Effectiveness of the Biopsychosocial Model-Based Exercise Approach (BETY) in Children and Adults Diagnosed With Scleroderma: A Single-Blind Randomized Controlled Trial
Brief Title: Investigating the Effectiveness of the Biopsychosocial Model-Based Exercise Approach in Children and Adults Diagnosed With Scleroderma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Orkun Tüfekçi, Principal Investigator, PT, PhD(c), Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FTREK25/154
Record Dates: First submitted 2025-12-06; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Scleroderma; Scleroderma, Localized; Scleroderma Systemic; Scleroderma (Limited and Diffuse); Systemic Sclerosis (SSc); Systemic Sclerosis - 2013 ACR/EULAR Classification Criteria; Juvenile Systemic Sclerosis
Keywords: biopsychosocial model; exercise; scleroderma; juvenile scleroderma
MeSH Terms: conditions — Scleroderma, Diffuse; Scleroderma, Localized; Scleroderma, Systemic; Juvenile systemic scleroderma; Motor Activity; Juvenile-onset scleroderma | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BETY session group (Experimental): Children and adults with scleroderma are participating in BETY sessions two times a week for 3 months.
  Interventions: Other: Cognitive Exercise Therapy Approach
- Control Group (Active Comparator): Children and adults with scleroderma are followed up with a home exercise program.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Cognitive Exercise Therapy Approach — The biopsychosocial model-based exercise approach (BETY) will be applied for 24 one-hour sessions, two days a week, for 3 months.
  Other Names: Bilişsel Egzersiz Terapi Yaklaşımı (BETY)
  Arms: BETY session group
Other: Control group — The control group will be followed up with a home exercise program, and notes will be taken.
  Arms: Control Group

SUMMARY:
This study aims to investigate the effectiveness of BETY, an exercise approach based on the biopsychosocial model, in children and adults diagnosed with scleroderma.

DETAILED DESCRIPTION:
EULAR recommendations on non-pharmacological treatment of scleroderma emphasize physical activity and patient education, disease-specific, evidence-based management strategies tailored to the individual, and self-management. Physical exercise is the most widely studied disease management strategy in scleroderma.

There is a reported need for biopsychosocial treatment approaches in disease management for cases and individuals diagnosed with scleroderma; therefore, the use of biopsychosocial approaches in the field of exercise is also recommended.

The Cognitive Exercise Therapy Approach (BETY), an innovative exercise approach developed for adults diagnosed with rheumatic diseases, also aims to promote behavioral change through exercises that provide pain management and functional gains in pediatric rheumatology, and to prevent social isolation through group support. As in adults, there is a need for exercise approaches, such as BETY, that align with the biopsychosocial model in pediatric cases.

BETY, previously implemented via telerehabilitation in individuals diagnosed with systemic sclerosis, has been shown to have beneficial effects on functionality, muscle strength, vascular structures, inflammatory markers, and biopsychosocial status.

In this context, there is a clear need for interventions that support both children and adults diagnosed with scleroderma physically and psychosocially. This study aims to investigate the effectiveness of BETY, an exercise approach based on the biopsychosocial model, in children and adults diagnosed with scleroderma.

ELIGIBILITY:
*For a child diagnosed with scleroderma*

Inclusion Criteria:

* Cases diagnosed with scleroderma,
* Cases aged 7-18 years will be included.

Exclusion Criteria:

* Advanced heart/lung/liver/kidney disease, neurological disease, and malignancies
* Cases that are not willing to participate in the study will be excluded.
* History of developmental delay
* Having participated in a regular exercise program for the past 3 months
* Individuals who are not willing to participate in the study

*For adults diagnosed with scleroderma*

Inclusion Criteria:

* Individuals diagnosed with scleroderma,
* Individuals over the age of 18 will be included.

Exclusion Criteria:

* Advanced heart/lung/liver/kidney disease, neurological disease, and malignancies
* Individuals who are not willing to participate in the study will be excluded.
* Having participated in a regular exercise program for the past 3 months
* Individuals who are not willing to participate in the study

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-12-04 (Actual); Primary Completion 2027-12-04 (Estimated); Study Completion 2027-12-04 (Estimated)

PRIMARY OUTCOMES:
Juvenile Arthritis Biopsychosocial Scale-JAB-Q-Patient | Six months
  It is a patient/parent-centered measurement method that helps assess the patient's biopsychosocial aspects, such as disease activity, posture, functional and psychosocial status, fatigue, and school performance. The results from the questions are used to assess the functional status of children, while their psychosocial status is recorded based on their answers to 21 questions (ranging from 0 to 358). A high score indicates a poor psychosocial status.
Cognitive Exercise Therapy Approach-Biopsychosocial Questionnaire (BETY-BQ) | Six months
  It was standardized as a biopsychosocial assessment tool and is scored using a 5-point Likert scale, with each item rated from 0 to 4 points. A high total score on the 30-item scale indicates a high level of biopsychosocial impact.
Modified Rodnan skin score (MRSS) | Six months
  A pediatric and adult rheumatologist assessed it. The MRSS evaluates skin thickening in 17 body regions, graded from 0 (normal) to 3 (severe skin thickening). The total score ranges from 0 to 51, with increased scores indicating poor skin involvement.
Localized Scleroderma Assessment Tool (LoSCAT) | Six months
  LoSCAT consists of two sections: the modified Localized Skin Severity Index, which measures disease activity, and the Localized Scleroderma Damage Index, which assesses damage (usually scored between 0 and 3). The Localized Skin Severity Index evaluates the color of the lesion border for erythema, skin thickness, and the presence of new lesions or lesion extension. In the Localized Scleroderma Damage Index, three areas of cutaneous damage are combined to obtain a score. These areas evaluate hyperpigmentation or hypopigmentation, whichever is more prominent, as well as dermal atrophy, subcutaneous atrophy, and dyspigmentation.
6-Minute Walk Test | Six months
  Participants are asked to walk as quickly as they can along a 30-meter corridor. The total distance will be measured in meters. Fatigue, pain, and dyspnea will be monitored using the Modified Borg Scale.

SECONDARY OUTCOMES:
Childhood Health Assessment Questionnaire (CHAQ) | Six months
  It assesses the functional abilities of children diagnosed with rheumatic diseases in their daily living activities. It consists of eight subscales (dressing and personal care, standing up, eating, walking, body care, reaching, grasping, activities) (0-3) and also assesses pain and general well-being using a visual analog scale (0-100). A high score indicates low functionality.
Juvenile Arthritis Quality of Life Questionnaire (JAQQ) | Six months
  It consists of 74 items covering various health domains, including physical functioning, emotional well-being, and general symptoms. The items are divided into four dimensions related to the child's quality of life: gross motor function (GMF), fine motor function (FMF), psychosocial function (PF), and systemic or general symptoms (SGS). Each domain is scored on a Likert-type scale from 1 to 7, with higher scores indicating poorer health-related quality of life. There is also a "not applicable to me" option for the items. The scale also includes a pain measurement (10 cm Visual Analog Scale (VAS)) to assess pain, but this score is not included in the total score.
Child and Adolescent Scale of Participation (CASP) | Six months
  It is a 20-question survey that assesses children's and adolescents' community participation in school, neighborhood, and local settings. The survey is divided into four sections: 6 questions about home participation, four questions about neighborhood and community involvement, five questions about school participation, and five questions about home and community engagement. It is rated on a scale of "expected for their age (full participation), somewhat limited, very limited, unable to participate, and inapplicable." The survey is completed by the child's family or primary caregiver. The person filling out the questionnaire is asked to select the answer that best describes the child's level of participation. The assessment is scored out of 100 points, with higher scores indicating greater participation.
Juvenile Arthritis Biopsychosocial Scale-JAB-Q-Family | Six months
  JAB-Q is a multidimensional questionnaire and a parent (family) form. Developed in Turkish by Ünal and colleagues, the questionnaire is completed by one of the child's parents. The family form evaluates the parents' biopsychosocial status from their own perspective and provides scores ranging from 0 to 102. Higher scores indicate a worse biopsychosocial status.
Pediatric Eating Assessment Scale (PEDI-EAT-10) | Six months
  It is used to evaluate swallowing disorders in pediatric patients. It was developed as the pediatric version of the EAT-10, which is used in adults. The PEDI-EAT-10 comprises 10 questions, each with a Likert scale ranging from 0 to 4 (0 = no problem, 4 = severe problem). The total score is calculated out of 40 points.
Pain Catastrophizing Scale-Parent (PCS-P) | Six months
  It is assessed using a 5-point Likert scale ranging from 0 (never) to 4 (always) and consists of 13 items. Similar to the child questionnaire, it assesses 3 domains: rumination, magnification, and helplessness. A total score between 0 and 52 is obtained; higher scores reflect a higher level of catastrophizing in parents.
Scleroderma Health Assessment Questionnaire (SHAQ) | Six months
  It was developed by adding five questions to the HAQ regarding Raynaud's phenomenon, digital ulcers, gastrointestinal, pulmonary, and general scleroderma symptoms, to be rated on a 15 cm line. The SHAQ total score ranges from 0 to 3. A high score indicates low functionality.
Short Form-36 (SF-36) | Six months
  It will be used to determine an individual's quality-of-life level. Each sub-parameter is scored between 0 and 100, with higher scores indicating better health status. The SF-36 scale has eight sub-parameters: general health perception, physical function, social function, pain, mental health, role difficulty due to physical reasons, role difficulty due to emotional reasons, and vitality. It contains 11 questions, each with 36 items.
Turkish Eating Assessment Tool (T-EAT-10) | Six months
  It is a questionnaire consisting of 10 questions with a Likert scale ranging from 0 to 4 (0 = no problem, 4 = severe problem). The total score is calculated out of 40 points by summing the responses given to each question. A score of 3 or higher is considered abnormal in the questionnaire.
Isokinetic Muscle Measurement | Six months
  Individuals' knee muscle strength will be assessed using the Biodex System 3 Pro® isokinetic device (Biodex Medical Systems Inc., Shirley, NY, USA), which is routinely used at Hacettepe University, Faculty of Medicine, Department of Sports Medicine. Before each assessment, participants will perform a 10-minute warm-up walk and then undergo maximal concentric isokinetic muscle strength tests of the knee flexors and extensors at angular velocities of 180°/s (10 repetitions) and 60°/s (5 repetitions), with 30-second rest intervals. Peak torque (PT) and average power (AP) will be recorded in newton-meters (Nm) and watts (W), respectively. Participants will be informed in advance of how to perform maximum-power training, and verbal encouragement will be provided during the tests.
Standard grip strength | Six months
  Hand grip strength will be evaluated using the Jamar hand dynamometer (Jamar; JLW Instruments, Chicago, IL), which is routinely used at Hacettepe University, Faculty of Medicine, Department of Sports Medicine. The test will be administered according to the American Hand Therapy Association's assessment recommendations. According to these recommendations, measurements will be taken with individuals seated in a chair without armrests, with the arm in adduction, the elbow at 90° flexion, the forearm in mid-rotation, and the wrist in a neutral position. A 15-second rest interval will be given between each measurement, and a total of three measurements will be taken. The average of the three scores will be recorded in kilograms-force.
Upper Extremity Proprioception Assessment | Six months
  Proprioception assessment will be performed at the wrist based on the principle of actively repeating a predetermined target angle. Measurements will be applied in all axes of movement of the wrist (flexion-extension, radial-ulnar deviation) on a surface showing a 180-degree angle range. Target angles are set at 30° for flexion-extension, 10° for radial deviation, and 15° for ulnar deviation.
Vascular Structures | Six months
  Vascular assessments will be performed using Doppler ultrasound in the Department of Radiology at Hacettepe University Faculty of Medicine. Spectral Doppler ultrasonography and shear wave elastography (SWE) measurements will be performed using a 9 MHz linear probe on a Siemens Acuson S2000 device.
  Doppler US measurements will be taken from the radial and posterior tibial arteries, and the Resistive Index (RI = peak systolic velocity - end-diastolic velocity/peak systolic velocity) value will be calculated. Three measurements will be taken from each artery, and the average RI value will be used.
  SWE measurements will be performed on the bilateral deltoid, rectus femoris, and forearm extensor muscles. Three measurements will be taken from the medial and lateral regions of each muscle, and the average SWE value will be obtained. Before all measurements, participants will rest for at least 30 minutes, and the probe will be placed parallel to the muscle fibers.
Inflammatory Markers | Six months
  Inflammatory markers will be collected via venipuncture during routine testing on the day of the clinical interview. Collected blood samples will be centrifuged at 2000 × g for 10 minutes and stored at -80 °C until kit analysis. Serum cytokine levels (TNF-α, IL-1, IL-6, IL-10) and serum irisin levels will be determined using ELISA kits.
Modified Hand Mobility in Scleroderma Test (mHAMIS) | Six months
  It is a functional test developed specifically for scleroderma to assess an individual's hand function. It evaluates four specific hand movements (finger flexion, finger extension, finger abduction, and dorsal extension). Scores range from 0 (normal) to 3 (complete failure) for each movement, with a total score ranging from 0 to 12.
Maximum mouth opening (MAO) | Six months
  After ensuring individuals open their mouths as widely as possible, the distance between the incisal edges of the central incisors in the upper and lower jaws is measured in millimeters and recorded.
Timed Up and Go Test | Six months
  The time it takes a person to rise from a chair with back support, walk 3 meters at a normal pace, and return to the chair is measured in seconds to evaluate lower-extremity balance. The test will be performed 3 times.
10-Step Stair Climbing Test | Six months
  To assess the subject's lower extremity strength and dynamic balance, the time taken to quickly climb and descend a staircase with 10 steps, each measuring 16-20 cm high and equipped with a handrail, is recorded in seconds. The test is repeated three times, and the times are recorded.
10-meter walk test | Six months
  The individual is on a 10-meter path. The assessment is performed in three repetitions and recorded in seconds.
30-second sit-to-stand test | Six months
  It is performed to evaluate lower-extremity endurance by having the individual stand up from a chair with their arms crossed over their chest, then sit back down. The individual is instructed to repeat this as quickly as possible for 30 seconds. The score for this assessment is the number of times the person fully rises from a seated position with arms crossed within 30 seconds.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Altındağ, Turkey (Türkiye)